CLINICAL TRIAL: NCT04574297
Title: The Impact of Genetic and Environmental Factors on the Progression of Chronic Pancreatitis：An Observational Study
Brief Title: An Observational Study on the Natural Course of Chronic Pancreatitis
Status: Active, not recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Principal Investigator, Changhai Hospital
Other Study IDs: CP-2011
Record Dates: First submitted 2020-09-27; First posted 2020-10-05 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pancreatitis; Genetic Mutation; Smoking, Tobacco; Drinking, Alcohol
MeSH Terms: conditions — Pancreatitis, Chronic; Tobacco Smoking; Alcohol Drinking | interventions — Smoking Devices; Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The remained peripheral blood sample after laboratory examinations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: smoking and alcohol assumption — documenting the change of smoking and drinking status during the follow-up period
Diagnostic Test: genetic sequencing — sequencing the susceptibility genes for CP, including serine protease inhibitor Kazal type 1, cationic trypsinogen, cystic fibrosis transmembrane conductance regulator, chymotrypsin C, etc.

SUMMARY:
To explore the impact on genetic and environmental factors for clinical manifestation, and the progression of chronic pancreatitis, including development of pancreatic insufficiency and other complications.

DETAILED DESCRIPTION:
The present study was an observational study aimed to explore the impact of genetic factors (rare pathogenic variants of CP) and environmental factors(smoking and alcohol assumption) on the clinical manifestation and progression of CP. The observation items included the pain patterns, incidence of complications of CP, pancreatic cancer and death.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of chronic pancreatitis
* agree to join the study and provide informed consent

Exclusion Criteria:

* autoimmune pancreatitis
* pancreatic cancer diagnosed within 2 years after the diagnosis of chronic pancreatitis
* the follow-up time less than 2 years
* patients presenting with diabetes and/or steatorrhea at onset of CP.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consequent patients with a diagnosis of CP in Changhai Hospital between 2010 to 2014
Sampling Method: Probability Sample
Enrollment: 798 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2030-12-31 (Estimated)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ru N, Xu XN, Cao Y, Zhu JH, Hu LH, Wu SY, Qian YY, Pan J, Zou WB, Li ZS, Liao Z. The Impacts of Genetic and Environmental Factors on the Progression of Chronic Pancreatitis. Clin Gastroenterol Hepatol. 2022 Jun;20(6):e1378-e1387. doi: 10.1016/j.cgh.2021.08.033. Epub 2021 Aug 28. PMID 34461303

RESULTS

PARTICIPANT FLOW:
Groups:
- G+/E+ Group: Genetic factor/s positive and environmental factor/s positive group. Patients with at least one rare pathogenic variant were considered genetic factor/s positive (denoted as G+). Patients with a history of either smoking or alcohol consumption were considered environmental factor/s positive (denoted as E+).
- G-/E+ Group: Genetic factor/s negative and environmental factor/s positive group.Patients with at least one rare pathogenic variant were considered genetic factor/s positive (denoted as G+). Patients with a history of either smoking or alcohol consumption were considered environmental factor/s positive (denoted as E+).
- G+/E- Group: Genetic factor/s positive group and environmental factor/s negative. Patients with at least one rare pathogenic variant were considered genetic factor/s positive (denoted as G+). Patients with a history of either smoking or alcohol consumption were considered environmental factor/s positive (denoted as E+).
- G-/E- Group: Genetic factor/s negative group and environmental factor/s negative. Patients with at least one rare pathogenic variant were considered genetic factor/s positive (denoted as G+). Patients with a history of either smoking or alcohol consumption were considered environmental factor/s positive (denoted as E+).
Period: Overall Study
Arm/Group | G+/E+ Group | G-/E+ Group | G+/E- Group | G-/E- Group
Started | 180 | 263 | 230 | 125
Completed | 180 | 263 | 230 | 125
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G+/E+ Group | G-/E+ Group | G+/E- Group | G-/E- Group | Total
Number analyzed (Participants) | 180 | 263 | 230 | 125 | 798
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.5 [29.0 to 43.0] | 44.0 [36.0 to 53.0] | 17.5 [12.0 to 29.8] | 36.0 [20.0 to 51.0] | 35.5 [21.3 to 46.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 147 | 81 | 239
  Male | 173 | 259 | 83 | 44 | 559
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 180 | 263 | 230 | 125 | 798
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 180 | 263 | 230 | 125 | 798

OUTCOME MEASURES:

1. Primary Outcome: the Number of Patients Developing Pancreatic Insufficiency
Description: The primary endpoint was the number of patients developing pancreatic insufficiency, categorised as 1) diabetes and steatorrhea, 2) diabetes only, or 3) steatorrhea only.
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | G+/E+ Group | G-/E+ Group | G+/E- Group | G-/E- Group
Number analyzed (Participants) | 180 | 263 | 230 | 125
Participants | 82 | 130 | 55 | 36

2. Secondary Outcome: Death
Description: all-cause death
Time Frame: 20 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 years.
Description: The definition of adverse event and/or serious adverse event is in accordance with the clinicaltrials.gov Definitions.
Groups:
- G+/E+ Group: genetic factor/s positive and environmental factor/s positive group Patients with at least one rare pathogenic variant were considered genetic factor/s positive (denoted as G+).
  Patients with a history of either smoking or alcohol consumption were considered environmental factor/s positive (denoted as E+).
- G-/E+ Group: genetic factor/s negative and environmental factor/s positive group Patients with at least one rare pathogenic variant were considered genetic factor/s positive (denoted as G+).
  Patients with a history of either smoking or alcohol consumption were considered environmental factor/s positive (denoted as E+).
- G+/E- Group: genetic factor/s positive group and environmental factor/s negative Patients with at least one rare pathogenic variant were considered genetic factor/s positive (denoted as G+).
  Patients with a history of either smoking or alcohol consumption were considered environmental factor/s positive (denoted as E+).
- G-/E- Group: genetic factor/s negative group and environmental factor/s negative
Arm/Group | G+/E+ Group | G-/E+ Group | G+/E- Group | G-/E- Group
All-Cause Mortality (participants affected / at risk) | 6/180 | 9/263 | 4/230 | 5/125
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/263 | 0/230 | 0/125
Other Adverse Events (participants affected / at risk) | 0/180 | 0/263 | 0/230 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT04574297/Prot_SAP_000.pdf